CLINICAL TRIAL: NCT02195466
Title: A Single Centre, Open-label Study, in Healthy Adult Volunteers, to Determine the Effects of Single-dose and Steady-state TPV/RTV 500/200 mg on the Steady-state Pharmacokinetics of Fluconazole 100 mg qd (200 mg Loading Dose)
Brief Title: Effects of Single-dose and Steady-state TPV/RTV on the Steady-state Pharmacokinetics of Fluconazole in Healthy Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1182.10
Record Dates: First submitted 2014-07-18; First posted 2014-07-21 (Estimated); Last update posted 2014-07-21 (Estimated); Status verified 2014-07

CONDITIONS: Healthy
MeSH Terms: interventions — tipranavir; Ritonavir; Fluconazole

ARMS (1):
- TPV + RTV + FCZ (Experimental)
  Interventions: Drug: Tipranavir (TPV); Drug: Ritonavir (RTV); Drug: Fluconazole (FCZ)

INTERVENTIONS:
Drug: Tipranavir (TPV) — 500 mg bid on days 7-14
Drug: Ritonavir (RTV) — 200 mg bid on days 7-14
Drug: Fluconazole (FCZ) — 200 mg loading dose on day 1, followed by 100 mg qd until day 13

SUMMARY:
Study to determine the effects of single-dose and steady-state TPV/RTV 500/200 mg on the steady-state pharmacokinetics of fluconazole

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects between 18 and 60 years of age inclusive
* A Body Mass Index (BMI) between 18 and 29 kg/m2
* Signed informed consent prior to trial participation
* Ability to swallow multiple large capsules without difficulty
* Acceptable laboratory values that indicate adequate baseline organ function are required at the time of screening. Laboratory values are considered to be acceptable if severity is less than or equal to Grade 1, based on the AIDS Clinical Trials Group (ACTG) Grading Scale. All abnormal laboratory values greater than Grade 1 are subject to approval by the trial clinical monitor
* Acceptable medical history, physical examination, 12-lead electrocardiogram, and chest X-ray (if not conducted within the last 12 months and deemed necessary by investigator) are required prior to entering the treatment phase of the study
* Willingness to abstain from the following starting 14 days prior to any administration of study drugs up until the end of the study:

  * Grapefruit or grapefruit juice
  * Red wine
  * Seville oranges
  * St. John's Wort or Milk Thistle
* Willingness to abstain from alcohol starting 2 days prior to administration study drug up to the end of the study
* Willingness to abstain from the following within 72 hours of pharmacokinetics (PK) sampling:

  * Garlic supplements
  * Methylxanthine containing drinks (coffee, tea, cola, energy drinks, chocolate, etc.)
* Willingness to abstain from over the counter herbal medications for the duration of the study
* Have been non-smokers for 3 months
* Willingness to abstain from vigorous physical exercise during intensive PK Days 6, 7, 13
* Reasonable probability for completion of the study

Exclusion Criteria:

* Female subjects who are of reproductive potential and:

  * Have a positive serum β-human chorionic gonadotropin (hCG) at Visit 1, or on Day 0 or Day 1
  * Have not been using a barrier contraceptive method for at least 3 months prior to Visit 3 (Day 1)
  * Are not willing to use a reliable method of barrier contraception (such as diaphragm with spermicidal cream/jelly or condoms with spermicidal foam), during the trial and 60 days after completion/termination
  * Are breast-feeding
* Participation in another trial with an investigational medicine within 60 days prior to Day 0 (Visit 2)
* Use of any prohibited medication listed in the protocol within 30 days prior to Day 0 (Visit 2)
* Use of any pharmacological contraceptive (including oral, patch or injectable contraceptives) within 1 month of study initiation and for the duration of the study. Use of Depo-Provera is excluded for six months prior to study initiation
* Use of hormone replacement therapy within 1 month of study initiation and for the duration of the study
* Administration of antibiotics within 10 days prior to Day 0 (Visit 2) or during the trial
* History of acute illness within the past 60 days. Subjects will be excluded for these disorders greater than sixty days if, in the opinion of the investigator, the subject does not qualify as a healthy volunteer
* History of thrombotic disease
* History of migraine headache
* Have serological evidence of hepatitis B virus (HBV) or hepatitis C virus (HCV)
* Have serological evidence of exposure to HIV
* Recent history of alcohol or substance abuse (within 1 year of study period)
* Blood or plasma donations within 30 days of Day 0 (Visit 2) or during the trial
* Subjects with a seated systolic blood pressure either <100 mm Hg or >150 mm Hg; resting heart rate either <50 beats/min or >90 beats/min. For subjects with a resting heart rate below 50, or above 90, the investigator may discuss exclusion with the medical monitor on a case-by-case basis
* Subjects with a history of any illness or allergy that, in the opinion of the investigator, might confound the results of the study or pose additional risk in administering TPV, RTV or FCZ to the subject
* Subjects who have had an acute illness within 2 weeks prior to Day 0 (Visit 2)
* Subjects who are currently taking any over-the-counter or prescription drug within 7 days prior to Day 0 (Visit 2) that, in the opinion of the investigator in consultation with the Boehringer Ingelheim (Canada) Ltd./Ltée clinical monitor, might interfere with either the absorption, distribution or metabolism of the test substances
* Known hypersensitivity to TPV, RTV, FCZ, or sulphonamide class of drugs
* Inability to adhere to the protocol
* Cautions or warnings in the FCZ package insert which, in the judgment of the investigator, should exclude a subject from the study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2003-06; Primary Completion 2003-07 (Actual)

PRIMARY OUTCOMES:
Area under plasma concentration time curve from 0-24 hours (AUC0-24h) for FCZ | up to 24 hours after administration of study drug
Maximum plasma concentration (Cmax) for FCZ | up to 24 hours after administration of study drug
Drug concentration in plasma at 24 hours after administration (Cp24h) for FCZ | up to 24 hours after administration of study drug

SECONDARY OUTCOMES:
AUC0-12h for TPV | up to 12 hours after administration of study drug
Cmax for TPV | up to 24 hours after administration of study drug
Drug concentration in plasma at 12 hours after administration (Cp12h) for TPV | up to 12 hours after administration of study drug
Oral clearance (Cl/F) for FCZ and TPV | up to 24 hours after administration of study drug
Time of maximum concentration (tmax) for FCZ and TPV | up to 24 hours after administration of study drug
Apparent terminal half life (t1/2) for FCZ and TPV | up to 24 hours after administration of study drug
Number of patients with adverse events | up to 6 weeks